CLINICAL TRIAL: NCT01939691
Title: Macular Edema Nepafenac vs. Difluprednate Uveitis Trial
Acronym: MEND
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty enrolling
Sponsor: University of California, San Francisco (Other)
Collaborators: Aravind Eye Hospitals, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-24978
Record Dates: First submitted 2013-09-06; First posted 2013-09-11 (Estimated); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Uveitis; Macular Edema
Keywords: difluprednate; prednisolone acetate; nepafenac
MeSH Terms: conditions — Uveitis; Macular Edema | interventions — difluprednate; nepafenac; prednisolone acetate

STUDY DESIGN:
Intervention Model Description: Randomized 3 arm (1:1:1) parallel design comparative effectiveness trial
Who Masked: Outcomes Assessor
Masking Description: Masked outcome assessment (evaluation of OCT and visual acuity)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Difluprednate (Experimental): Difluprednate 0.05% ophthalmic emulsion 4 times a day until Week 4, then decrease according to protocol (if resolution of edema at 4 weeks, decrease to 1 drop per day until Week 6, then stop; if not resolved, continue at 4 times a day until 6 weeks and then decrease to 1 drop per day until Week 8 if resolved, then stop). If macular edema not resolved (or reoccurs) by Week 8, treat per best medical judgement.
  Interventions: Drug: Difluprednate
- Nepafenac plus Prednisolone acetate (Experimental): Nepafenac 0.1% 3 times a day until resolution; prednisolone acetate 1% 4 times a day until Week 4, then decrease according to protocol (if resolution of edema at Week 4, decrease to 1 drop per day until Week 6, then stop; if not resolved, continue at 4 times a day until Week 6, then decrease to 1 drop per day until Week 8, then stop). If macular edema not resolved (or reoccurs) by Week 8, treat per best medical judgement.
  Interventions: Drug: Nepafenac; Drug: Prednisolone acetate
- Difluprednate plus Nepafenac (Experimental): Nepafenac 0.1% 3 times a day until resolution; Difluprednate 0.05% ophthalmic emulsion 4 times a day until Week 4, then decrease according to protocol (if resolution of edema at 4 weeks, decrease to 1 drop per day until Week 6, then stop; if not resolved, continue at 4 times a day until 6 weeks and then decrease to 1 drop per day until Week 8 if resolved, then stop). If macular edema not resolved (or reoccurs) by Week 8, treat per best medical judgement.
  Interventions: Drug: Difluprednate; Drug: Nepafenac

INTERVENTIONS:
Drug: Difluprednate — Difluprednate 0.05% - corticosteroid eyedrop
  Other Names: Durezol
  Arms: Difluprednate; Difluprednate plus Nepafenac
Drug: Nepafenac — Nepafenac 0.1% - NSAID eyedrop
  Other Names: Nevanac
  Arms: Difluprednate plus Nepafenac; Nepafenac plus Prednisolone acetate
Drug: Prednisolone acetate — prednisolone acetate 1% - corticosteroid eyedrop
  Other Names: Pred Forte, Econo Pred
  Arms: Nepafenac plus Prednisolone acetate

SUMMARY:
Macular edema is a condition in which there is swelling in the macula, the part of the retina that gives you your best vision. This swelling can cause your vision to decline. When diagnosed early and treated, you vision usually can be preserved. However, if the swelling goes untreated for a long time, it can cause permanent vision loss.

We think that the three eye drop regimens in this study, difluprednate, difluprednate plus nepafenac, and prednisolone acetate plus nepafenac, might be effective in treating uveitic macular edema. Patients who enter this study are randomized to one of the three regimens and followed for 24 weeks.

DETAILED DESCRIPTION:
Trial: Randomized 3 arm (1:1:1) parallel design comparative effectiveness trial

Stratification: Systemic corticosteroid/immunosuppressive therapy vs. none

Treatments: 1) difluprednate 0.05% 2) combination therapy of prednisolone acetate 1% with nepafenac 0.1% 3) combination therapy of difluprednate 0.05% with nepafenac 0.1%

Masking: Unmasked treatment administration; masked outcome assessment (evaluation of OCT and visual acuity)

Follow-up: 2, 4, 6, 8, and 24 weeks

Treatment protocol:

Patients will be randomized at enrollment to either:

* difluprednate 0.05% 4 drops per day
* prednisolone acetate 1% 4 drops per day and nepafenac 0.1% 3 drops per day
* difluprednate 0.05% 4 drops per day and nepafenac 0.1% 3 drops per day

If macular edema has not resolved at Week 4, continue study treatment at the same dose until Week 6.

If macular edema has resolved at Week 4, reduce study treatment as follows:

* difluprednate 0.05% 1 drop per day until Week 6, then stop
* prednisolone acetate 1% 1 drop per day and nepafenac 0.1% 3 drops per day until Week 6, then stop
* difluprednate 0.05% 1 drop per day and nepafenac 0.1% 3 drops per day until Week 6, then stop

If macular edema does not resolve at Week 4 but has resolved at Week 6, reduce study treatment at Week 6 as follows:

* difluprednate 0.05% 1 drop per day until Week 8, then stop
* prednisolone acetate 1% 1 drop per day and nepafenac 0.1% 3 drops per day until Week 8, then stop
* difluprednate 0.05% 1 drop per day and nepafenac 0.1% 3 drops per day until Week 8, then stop If macular edema resolves at Week 4 but reoccurs at Week 6, treat per best medical judgement.

After Week 8, there are no restrictions on the treatments patients may receive, and medications can be tapered further, discontinued, or changed at the discretion of the treating physician and patient preference. If a patient with previously resolved macular edema has a recurrence, the physician may treat according to best medical judgement.

ELIGIBILITY:
108 patients with uveitic ME will be enrolled at Aravind Eye Hospital in Madurai, India based on the following eligibility criteria:

Patient-level Inclusion criteria:

* ≥18 years of age
* Diagnosis of anterior, intermediate, posterior, or panuveitis (can be infectious or non-infectious)
* Inactive or minimally active inflammation according to Standardization of Uveitis Nomenclature criteria (≤ 0.5+ Anterior Chamber (AC) cells, ≤ 0.5+ vitreous haze and no active retinal/choroidal lesions)
* If on oral corticosteroids, a stable dose of <10 mg prednisone/day for >4 weeks
* If on systemic corticosteroid-sparing immunomodulatory therapy, a stable dose for >4 weeks
* If using prednisolone acetate 1% drops, stable regimen of ≤2 drops per day for >4 weeks
* If infectious uveitis, inflammation must be inactive or minimally active per definition above and on stable dose of treatment for ≥4 weeks with no anticipated changes to treatment during the trial

Eye-level Inclusion Criteria

* ME defined as thickening of the 1mm central subfield of the macula greater than 2 standard deviations above normal thickness (>320 µm by Heidelberg spectral-domain OCT) with or without the presence of intraretinal cysts.
* Baseline intraocular pressure >5 mmHg and <21 mmHg (current use ≤3 intraocular pressure-lowering medications and/or prior glaucoma surgery are acceptable)
* Media clarity and pupillary dilation sufficient to allow OCT testing and retinal photography
* Best-corrected visual acuity of 5/200 or better

Patient-level Exclusion Criteria

* Use of oral acetazolamide or other systemic carbonic anhydrase inhibitors at baseline
* Known allergy or hypersensitivity to any component of the study drugs
* Women who are pregnant or breastfeeding (pregnancy test should be administered prior to baseline fluorescein angiogram)
* Patients unwilling or unable to not wear contact lenses during the study period
* History of central serous chorioretinopathy in either eye

Eye-level Exclusion Criteria

* Intravitreal or periocular corticosteroid injection in the past 8 weeks, dexamethasone implant in the past 12 months, or a fluocinolone acetonide implant in the past 3 years
* Presence of an epiretinal membrane-noted clinically or by OCT-in the study eye, thought to be significant enough to preclude improvement of ME
* Previous pars plana vitrectomy
* History of severe glaucoma (C/D ratio > 0.9 or any notching of optic nerve to rim)
* Prior use of difluprednate or nepafenac in the past 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-09-12 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Central subfield thickness | 4 weeks
  Central subfield thickness measured by spectral domain optical coherence tomography adjusting for baseline thickness

SECONDARY OUTCOMES:
Resolution | 4 weeks
  proportion of patients with resolution of macular edema
Improvement | 4 weeks
  proportion of patients with improvement in macular edema defined as 20% or greater reduction in central subfield thickness by OCT or resolution of edema
recurrence | 4 weeks
  proportion of patients with recurrence of macular edema defined as greater than 20% increase in central subfield thickness to a value >320 microns by OCT or presence of cysts in an eye that previously had resolution of macular edema
Intraocular pressure (IOP) increase | 4 weeks
  number of patients with intraocular pressure increase at least 10mmHg over baseline
High IOP | 4 weeks
  Number of patients experiencing high intraocular pressure (> 24 mmHg)
Visual acuity | 4 weeks
  best-corrected visual acuity (ETDRS protocol)

CONTACTS AND LOCATIONS:
Overall Officials: Nisha Acharya, MD MS, Principal Investigator — University of California, San Francisco
Locations (3):
- India (3):
  - Aravind Eye Hospital, Coimbatore, Tamil Nadu
  - Aravind Eye Hospital, Madurai, Tamil Nadu
  - Aravind Eye Hospital, Pondicherry, Tamil Nadu

IPD SHARING:
Plan to Share IPD: No